CLINICAL TRIAL: NCT02786368
Title: Scale up of Enhanced Homestead Food Production for Improved Household Food Security and Nutrition in Cambodia
Brief Title: Scale up of Enhanced Homestead Food Production in Cambodia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Helen Keller International (Other); International Development Research Centre, Canada (Other Government)
Responsible Party: Principal Investigator, Tim Green, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H15-00720
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Food Supply
Keywords: Food Production; Inadequacy; Dietary zinc; Iron; vitamin A
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): For year one, this arm will receive no intervention. Usual agriculture production and income will be assessed monthly for one year. Additionally, every season (twice yearly), household food security and usual dietary intake of woman of reproductive age (WRA) and their child aged 6-59 mo will also be collected. After one year of implementation, this group will be offered the Enhanced Homestead Food Production package fully subsidized, as well as training on nutrition, WASH, gender and business/marketing.
  Interventions: Behavioral: Control group
- EHFP group (Experimental): Households will receive training and inputs for an Enhanced Homestead Food Production (EHFP) package. Participants will also receive educational components through inter-personal behavioural change communication on nutrition (Essential Nutrition Actions), Water Sanitation and Hygiene (WASH), gender, and business/marketing.
  Interventions: Behavioral: EHFP group

INTERVENTIONS:
Behavioral: Control group — A comparison group; no intervention for year 1, EHFP after 1 year of program implementation.
  Arms: Control group
Behavioral: EHFP group — Intervention group: training; inputs cost-sharing for EHFP activities.
  Arms: EHFP group

SUMMARY:
This project is a delayed pragmatic delayed-intervention cluster randomized control study in a subset of households (n=600) enrolled in a larger scale up program of enhanced homestead food production (EHFP) in Cambodia. The trial is designed to evaluate the impact of EHFP (home gardens only; home garden and fishponds; home gardens and poultry) versus control group on dietary intake of women and youngest child, household food security, income, and production throughout the agricultural cycle. Following administration of the baseline survey 300 households will be randomized to the EHFP package of their choosing (Intervention Group) for two years. The other 300 households will not receive any intervention during the first year and will act as the control group; data will be collected monthly on production and income generated from gardening (and other homestead food production activities) and at two points throughout the year 24-hour dietary recall data will be collected from the women head of the household (aged 15-49y) and the youngest child between the ages of 6 - 59 months. After one year, the control group will be offered the intervention (EHFP package of their choice) fully subsidized and the project team will collect identical data on intervention group for one year as described for the control group.

DETAILED DESCRIPTION:
Cambodia's economy has improved remarkably in the last decade, yet 80% of households experience some form of poverty, and 20% are severely impoverished. Food insecurity and its sequelae remain a problem, especially among rural farmers. As a solution Helen Keller International (HKI) implements a Enhanced Homestead Food Production (EHFP) model in Cambodia. EHFP, focusing on women farmers, fosters year-round environmentally sustainable production of nutrient-rich fruits, vegetables and animal-source foods. The program provides initial farming inputs coupled with technical assistance, nutrition education, and training on marketing and gender equity.

In 2012, HKI together with the University of British Columbia (UBC), conducted a 22-month randomized control trial of EHFP, known as 'Fish on Farms'. Using HKI's approach, 900 women farmers were randomized to three groups: 1) plant-based EHFP; 2) EHFP plus fishponds; or 3) a control. Remarkably, in less than two years working with women farmers, Fish on Farms established 300 fishponds and 600 gardens. In the fishponds, small nutrient-rich fish were raised for household consumption and larger fish were raised for consumption or sale. After two years, households in both EHFP arms saw improvements in food production, income generation, food security, dietary diversity, and dietary intake of certain micronutrients relative to the control. However, the randomized-control trial (RCT) approach did have a number of issues, and gaps that need to be addressed were identified. Attrition was high, perhaps in part because of better opportunities for women, but also because women were not given a choice in the type of HFP activity to participate in. Further, the project provided many inputs for free so the women were not as invested as they might have otherwise been. Other issues identified were a lack of market access for sale of produce and fish, gender inequities, and a need to better capture the seasonality of food production and consumption at the household level.

Building on lessons learned from the pilot study (Fish on Farms), this pragmatic delayed-intervention cluster randomized control study includes rigorous monitoring of production throughout the agricultural cycle as well as multiple 24-hour dietary recalls with improved methodology and frequency to better capture dietary intake. Women are self-selecting to participate, and are provided access to micro-credit institutions or other cost-sharing options so that women have a greater financial stake in EHFP leading to more successful farmers. Participants will also able to select from more EHFP options that include home gardens, poultry and fish.

The ultimate goal of the program is to provide evidence of an integrated model of EHFP that has scalability and sustainability to improve the livelihoods of Cambodians and possibly the larger region.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (15-49 y)
* Child aged 6 - 59 months
* Demonstrate a willingness to cost-share on EHFP inputs
* Have suitable land for Enhanced Homestead Food Production activities

Exclusion Criteria:

* Not meeting the above inclusion criteria

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1318 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Difference in mean intake of zinc | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Sample size was calculated to detect a difference in zinc and vitamin A intake between any two groups, with 80% power and alpha of 0.05, assuming a 30% attrition. Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean intake of vitamin A | Measurements will be made for women of reproductive age aand the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Sample size was calculated to detect a difference in zinc and vitamin A intake between any two groups, with 80% power and alpha of 0.05, assuming a 30% attrition. Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.

SECONDARY OUTCOMES:
Household food security | Baseline (2016) through to study completion, on average 2 years
  Measured with a questionnaire to calculate the Household Food Insecurity Access Scale score. Unit: percentage of households.
Women's empowerment / gender equity | Baseline (2016) through to study completion, on average 2 years
  Measured by questionnaire using the Women's Empowerment in Agriculture Index (WEAI) household decision-making on production and use of money modules. Percentage of women over a calculated score.
Incremental net monetary benefit | Monthly for 1 year
  The economic evaluation of the program will take the form of a cost-benefit analysis from the perspective of the project. Costs will be determined from HKI's budget sheets and input use (resource use) reported by study participants monthly. Benefits will be measured in terms of total kilograms of each variety of food produced over a 12 month period (collected every month) and monetized using local market values that are collected every month.
WASH practices | Baseline (2016) through to study completion, on average 2 years
  Using questionnaire on knowledge, percentage of women giving adequate answer.
Difference in mean energy intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean protein intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean fat intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean riboflavin intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean thiamin intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.
Difference in mean iron intake | Measurements will be made for women of reproductive age and the youngest child in the household (> 6 mo < 60 mo) at baseline and ~ 7 months later
  Measured by 24 hour dietary recall surveys with repeat recalls on a sub-set of the sample in order to adjust for intra-individual variations in intake and provide an estimate of usual intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Timothy D Green, Vancouver, British Columbia, Canada